CLINICAL TRIAL: NCT00293436
Title: A Phase I/II Study of Celecoxib and Erlotinib Hydrochloride as Adjuvant Therapy for High Risk Patients With a History of Hepatocellular Carcinoma
Brief Title: Celecoxib and Erlotinib in Treating Patients With Liver Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000458055; UCSF-04459; UCSF-H43059-26066-02
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized resectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Celecoxib; Erlotinib Hydrochloride; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: celecoxib
Drug: erlotinib hydrochloride
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Celecoxib and erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. Celecoxib may also stop the growth of liver cancer by blocking blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving celecoxib together with erlotinib and to see how well they work in treating patients with liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of adjuvant celecoxib and erlotinib hydrochloride for patients with hepatocellular carcinoma (HCC) at high risk for recurrence. (phase I)
* Assess disease-free and overall survival of patients treated with adjuvant celecoxib and erlotinib hydrochloride. (phase II)

Secondary

* Determine the maximum tolerated dose of celecoxib and erlotinib hydrochloride for the phase II portion of this trial. (phase I)

OUTLINE: This is a phase I, dose-escalation study followed by an open-label, phase II study. Patients are assigned to a treatment according to Child-Pugh class of cirrhosis (class A/noncirrhotic vs class B).

* Phase I: Patients receive oral celecoxib once or twice daily and oral erlotinib hydrochloride once daily. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of celecoxib and erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Separate dose escalations are conducted in the 2 groups according to liver dysfunction.

* Phase II: Patients receive celecoxib and erlotinib hydrochloride as in phase I at the MTD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological evidence of hepatocellular carcinoma (HCC)

  * No evidence of residual or recurrent disease
* Received 1 of the following therapies:

  * Tumor resection between 4-8 weeks prior to study enrollment
  * Transarterial chemo-embolization between the past 4-8 weeks
  * Radiofrequency ablation and percutaneous ethanol injection (sequential or combinations thereof) between the past 2-8 weeks
* Meets 1 of the following high-risk features for recurrence:

  * History of resection of a single HCC > 5 cm
  * History of multifocal HCC (includes microsatellite disease found at time of resection)
  * History of vascular invasion (macro or micro)
  * History of poorly differentiated HCC
  * Underlying cirrhosis
* No Child-Pugh class C cirrhosis

PATIENT CHARACTERISTICS:

* Absolute neutrophil count > 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.0 mg/dL
* AST/ALT ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* INR ≤ 1.5 times ULN
* Albumin ≥ 2.5 g/dL
* ECOG performance status 0-2
* Life expectancy ≥ 2 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after completion of study treatment
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* Patients must agree not to wear contact lenses
* No history of ulcer disease or gastrointestinal bleeding
* No myocardial infarction within the past 18 months
* No cerebral vascular event within the past 18 months
* No history of aspirin or NSAID-induced asthma
* No history of Gilbert's syndrome
* No history of hypersensitivity reaction or allergy to sulfa drugs, aspirin, or other NSAIDs
* No liver transplantation candidates for phase I portion of the study
* No New York Heart Association class III or IV cardiac disease
* No interstitial lung disease
* No gastrointestinal disease prohibiting oral medication or requiring IV alimentation
* No active peptic ulcer disease
* No unstable angina pectoris
* No ongoing, active, or untreated infection
* No hypersensitivity to celecoxib
* No rising alpha-fetal protein (AFP) not attributable to hepatitis B or C virus
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* No prior liver transplantation
* No prior chemotherapy or biologic therapy in the adjuvant setting
* No prior chest or mantle radiotherapy
* No concurrent aspirin or other nonsteroidal anti-inflammatory drug (NSAID)
* No concurrent interferon
* No concurrent oral steroids
* No concurrent anticoagulant therapy
* No concurrent CYP3A4 inducers or inhibitors
* No concurrent commercial or other investigational anticancer agents or therapies
* No concurrent selective cyclooxygenase-2 inhibitors
* No concurrent antineoplastic or antitumor agents, including chemotherapy, radiotherapy, immunotherapy, or hormonal anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01

PRIMARY OUTCOMES:
Safety (phase I)
Disease-free survival (phase II)

SECONDARY OUTCOMES:
Maximum tolerated dose (phase I)
Overall survival (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Alan P. Venook, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States